CLINICAL TRIAL: NCT06384898
Title: Remote Tai Chi for Knee Osteoarthritis: An Embedded Pragmatic Trial
Brief Title: Remote Tai Chi for Knee Osteoarthritis
Acronym: TAICHIKNEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Boston Medical Center (Other); University of California, Los Angeles (Other); The Cleveland Clinic (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002259; UH3AT012413 (NIH)
Record Dates: First submitted 2024-03-26; First posted 2024-04-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Pragmatic Clinical Trial; Implementation Science; Mind-body Therapies; Tai Chi; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The study is an individually randomized group-treatment (IRGT) trial. Individuals randomly allocated to remote Tai Chi receive the intervention with other participants through an instructor.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi + Routine Care (Experimental): The intervention will be delivered via a HIPAA-secure web-based video platform. All remote Tai Chi sessions will be 60 minutes, twice a week, for 3 months. All program components will use the Yang style Tai Chi, and every session will include warm up, review of principles, meditation with movement, breathing techniques and relaxation.
  Interventions: Other: Remote Tai Chi
- Routine Care (No Intervention): Participants will be encouraged to continue their ongoing care for Knee OA by their providers. In addition, primary care providers and other participating clinicians in the health system will receive information from the study team on routine care or "2019 ACR Guideline-Based Care." At the end of the 12-month trial period, routine care participants will be offered access to recordings for the full 3-month Tai Chi program (24 sessions).

INTERVENTIONS:
Other: Remote Tai Chi — Tai Chi mind-body exercise is a complex, multi-component nonpharmacological intervention integrating physical, psychological, emotional, and behavioral elements.
  Arms: Tai Chi + Routine Care

SUMMARY:
The goal of this pragmatic randomized trial is to evaluate the effectiveness of remote Tai Chi to treat knee pain in adults with knee osteoarthritis. The main questions the trial aims to answer are:

* Compared to routine care, will patients with Knee OA receiving remote Tai Chi exhibit greater improvement in knee-related pain (WOMAC pain score, primary outcome), pain interference (PROMIS-Pain Interference, secondary outcome), and health-related quality of life at 3 months?
* Does remote tai chi decreases healthcare utilization and analgesic use over the one-year study period?

Researchers will compare remote Tai Chi added to routine care to routine care alone to see if remote tai chi works to treat knee osteoarthritis pain. Participants will participate in remotely delivered web-based tai chi sessions, twice a week for 12 weeks, or will continue to receive routine care. Participants will be followed for 12 months after randomization.

DETAILED DESCRIPTION:
Investigators will conduct a 12-month embedded, pragmatic, hybrid type 1 effectiveness-implementation, individually randomized group-treatment trial that will compare the effects of a 3-month twice weekly remotely delivered web-based Tai Chi intervention plus routine care versus routine care alone across four health care systems (Tufts Medical Center, Boston Medical Center, University of California Los Angeles Health, and Cleveland Clinic) in four geographic regions (Eastern Massachusetts, Southern California, Northeast Ohio (Cleveland Clinic), Southern Florida (Cleveland Clinic). Investigators will enroll a total of 480 diverse patients with a clinical diagnosis of Knee OA. Participants will be evaluated at baseline and 3 months, with additional follow-up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Treating clinician diagnosis of knee osteoarthritis
* Have a score of 40 (visual analog version) or greater on at least 1 of the 5 questions in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale (range of 0 to 100, with higher scores indicating greater pain) at baseline.
* Able to provide informed consent
* If randomized to the Routine Care group, willing to abstain from Tai Chi programs until completion of the study
* If randomized to the Tai Chi group, willing to comply with the Tai Chi program (twice-a-week remote sessions for 12 weeks)
* Has access to a home computer or device that will allow telehealth (bidirectional audio and video) delivery of the intervention
* Is an active patient at one of the 4 participating healthcare system

Exclusion Criteria:

* Currently practicing Tai Chi
* Serious medical conditions (e.g., dementia, significant neurological deficits or neurodegenerative disorder, active cancer treatment, psychosis, sensory deficits) limiting the participant's ability to participate in the Tai Chi safely, as determined by the principal investigators
* Unable to walk without a cane or other assistive device
* Any previous or scheduled knee replacement
* Reports severe depression defined by a Beck Depression Inventory (BDI-II) score of 29 or more.
* Reports suicidal ideations defined by a score on BDI-II item of 2 or 3 ('I would like to kill myself' or 'I would kill myself if I had the chance').
* Not English speaking
* Enrollment in any other clinical trial within the last 30 days

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC Pain Score | 3 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score rated on a Visual Analog Scale (VAS) of 0-100 mm.

SECONDARY OUTCOMES:
PROMIS Pain Interference score | 3 months from randomization
  The PROMIS Pain Interference short form 6b evaluates the extent to which pain interferes with physical, emotional and social activities. The raw score ranges between 6-30 and the T score ranges between 41.0-78.3, with higher scores indicating that pain has a greater negative impact.
SF-12 PCS score | 3 months from randomization
  The 12-item Short Form Health Survey (SF-12) has two summary scales, the Mental Health Component Score (MCS) and the Physical Component Score (PCS). Both scores range from 0 to 100, with higher scores indicating better mental and physical health.
Number of knee joint injections | 12 months from randomization
  Total number of intra-articular injections identified through EHR and patient questionnaires.

OTHER OUTCOMES:
WOMAC Pain Score | 6 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC Pain Score | 12 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score rated on a Visual Analog Scale (VAS) of 0-100 mm.
PROMIS Pain Interference score | 6 months from randomization
  The PROMIS Pain Interference short form 6b evaluates the extent to which pain interferes with physical, emotional and social activities. The raw score ranges between 6-30 and the T score ranges between 41.0-78.3, with higher scores indicating that pain has a greater negative impact.
PROMIS Pain Interference score | 12 months from randomization
  The PROMIS Pain Interference short form 6b evaluates the extent to which pain interferes with physical, emotional and social activities. The raw score ranges between 6-30 and the T score ranges between 41.0-78.3, with higher scores indicating that pain has a greater negative impact.
SF-12 PCS score | 6 months from randomization
  The 12-item Short Form Health Survey (SF-12) has two summary scales, the Mental Health Component Score (MCS) and the Physical Component Score (PCS). Both scores range from 0 to 100, with higher scores indicating better mental and physical health.
SF-12 PCS score | 12 months from randomization
  The 12-item Short Form Health Survey (SF-12) has two summary scales, the Mental Health Component Score (MCS) and the Physical Component Score (PCS). Both scores range from 0 to 100, with higher scores indicating better mental and physical health.
WOMAC total score | 3 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score calculated by summing the pain, stiffness, and physical function subscales, rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC total score | 6 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score calculated by summing the pain, stiffness, and physical function subscales, rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC total score | 12 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score calculated by summing the pain, stiffness, and physical function subscales, rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC Pain Score on nominated activity chosen at baseline | 3 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score rated on a Visual Analog Scale (VAS) of 0-100 mm.(Considering ALL the ways Knee PAIN affects participants, which activity is most important to participants today?)
WOMAC Pain Score on nominated activity chosen at baseline | 6 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score rated on a Visual Analog Scale (VAS) of 0-100 mm.(Considering ALL the ways Knee PAIN affects participants, which activity is most important to participants today?)
WOMAC Pain Score on nominated activity chosen at baseline | 12 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score rated on a Visual Analog Scale (VAS) of 0-100 mm.(Considering ALL the ways Knee PAIN affects participants, which activity is most important to participants today?)
WOMAC function score | 3 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function score rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC function score | 6 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function score rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC function score | 12 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function score rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC stiffness score | 3 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness score rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC stiffness score | 6 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness score rated on a Visual Analog Scale (VAS) of 0-100 mm.
WOMAC stiffness score | 12 months from randomization
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness score rated on a Visual Analog Scale (VAS) of 0-100 mm.
Patient's global assessment score | 3 months from randomization
  VAS 0-100
Patient's global assessment score | 6 months from randomization
  VAS 0-100
Patient's global assessment score | 12 months from randomization
  VAS 0-100
PROMIS sleep disturbance OA Knee- Short Form 6a | 3 months from randomization
  PROMIS sleep disturbance OA knee raw score ranges between 6-30 and the T score ranges between 29.8-76.1, with higher scores indicates greater sleep disturbance.
PROMIS sleep disturbance OA Knee- Short Form 6a | 6 months from randomization
  PROMIS sleep disturbance OA knee raw score ranges between 6-30 and the T score ranges between 29.8-76.1, with higher scores indicates greater sleep disturbance.
PROMIS sleep disturbance OA Knee- Short Form 6a | 12 months from randomization
  PROMIS sleep disturbance OA knee raw score ranges between 6-30 and the T score ranges between 29.8-76.1, with higher scores indicates greater sleep disturbance.
Beck Depression Inventory-II score | 3 months from randomization
  The Beck Depression Inventory-II score ranges between 0-63, with higher scores indicating more severe depression symptoms.
Beck Depression Inventory-II score | 6 months from randomization
  The Beck Depression Inventory-II score ranges between 0-63, with higher scores indicating more severe depression symptoms.
Beck Depression Inventory-II score | 12 months from randomization
  The Beck Depression Inventory-II score ranges between 0-63, with higher scores indicating more severe depression symptoms.
SF-12 MCS score | 3 months from randomization
  The SF-12 Mental Component Score ranges between 0-100.
SF-12 MCS score | 6 months from randomization
  The SF-12 Mental Component Score ranges between 0-100.
SF-12 MCS score | 12 months from randomization
  The SF-12 Mental Component Score ranges between 0-100.
OMERACT/OARSI responder | 3 months from randomization
  Number of participants who meet the OMERACT/OARSI responder criteria
OMERACT/OARSI responder | 6 months from randomization
  Number of participants who meet the OMERACT/OARSI responder criteria
OMERACT/OARSI responder | 12 months from randomization
  Number of participants who meet the OMERACT/OARSI responder criteria
Receipt of knee surgery | 12 months from randomization
  Number of Participants who receive knee surgery.
Pain medication use | 3 months from randomization
Pain medication use | 6 months from randomization
Pain medication use | 12 months from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts Medical Center; Robert Saper, MD, MPH, Principal Investigator — The Cleveland Clinic; Eric Roseen, DC, PhD, Principal Investigator — Boston Medical Center; Helen Lavetrsky, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit and share de-identified individual patient data as described in our Data Management and Sharing Plan and will follow NIH policies for data sharing
Supporting Information: Study Protocol, SAP
Time Frame: The time of results publication or the end of the funding period.

REFERENCES:
- See also: Study website — https://sites.tufts.edu/taichiknee/